CLINICAL TRIAL: NCT06288399
Title: Prevalence and Economic Burden of Obesity-related Comorbidities in the Gulf Region: A Retrospective, Observational Study
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7688; U1111-1292-7248 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Obesity Group: Adults with diagnosis of obesity and obesity-related comorbidities
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The aim of this study is to assess the annual prevalence of ORCs among adult people with obesity in the real-world clinical setting across the Gulf region. In addition, the study will describe the annual HCRU and associated costs of obesity and ORCs, describe the demographics and clinical characteristics of adult people with obesity, as well as estimate the annual incidence and point prevalence of the ORCs among adult people with obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Local national (male or female) of Arab ethnicity, age above or equal to 18 years at index date
2. Primary or secondary diagnosis of obesity (BMI above or equal to 30 kg/m2) at index date
3. Minimum of 1 visit with BMI recorded between months 1 and 6 following index date, and minimum of 1 visit with BMI recorded between months 7 and 12 following index date.

There should be a minimum time gap of 3 months between the BMI records and the BMI must be above or equal 30 kg/m2 at each visit. If there are multiple visits during the 12-month observation period, then a mean BMI above or equal 30 kg/m2 must be maintained during the observation period.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having collected data of the participants in this study already.
2. Participation in an interventional trial during the 12-month observation period
3. Conditions associated with unintentional weight change
4. Participants who underwent bariatric surgery within 18 months prior to the index date
5. Participants with non-ambulatory disability diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with diagnosis of obesity and obesity-related comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 1316 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of Obesity Related Comorbidities (ORC, existing/newly diagnosed) among adult people with obesity (BMI above or equal to 30 kg/m2) over a period of 12 months across the Gulf region in primary and secondary hospitals as well as obesity clinics | 12-month observation period from the index date (Day 1) to Month 12 after the index date (+12 months)
  Percentage (and 95% CI)
  ORC: Dyslipidaemia, Hypertensive diseases, Type 2 diabetes mellitus, Non-alcoholic fatty liver disease, Coronary artery disease

CONTACTS AND LOCATIONS:
Locations (7):
- Kuwait (3):
  - Farwaniya Hospital, Farwaniya
  - Al-Adan Hospital, Hadiya
  - Al-Amiri Hospital, Kuwait City
- Oman (2):
  - National Diabetes and Endocrine Center, Muscat
  - Samail Polyclinic, Samail
- Qatar (2):
  - Hamad General Hospital, Doha
  - PHCC, Doha

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com